CLINICAL TRIAL: NCT05521217
Title: Quantification of the Postural Muscles Mechanical Properties of Individuals With Spinal Muscular Atrophy Using Myotonometer: Intra- and Inter Examiner Reliability
Brief Title: Myotonometer Intra- and Inter Examiner Reliability on Spinal Muscular Atrophy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-10840098-772.02-3771
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-08

CONDITIONS: Muscle Tone Poor; Spinal Muscular Atrophy
MeSH Terms: conditions — Muscle Hypotonia; Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Spinal Muscular Atrophy: The patients were included if they were between 0 to 4 yeats, with a diagnosis of Spinal Muscular Atrophy.
  Interventions: Diagnostic Test: MyotonPRO
- Healthy children: The healthy age-matched control group was included.
  Interventions: Diagnostic Test: MyotonPRO

INTERVENTIONS:
Diagnostic Test: MyotonPRO — Evaluation of biomechanics and viscoelastic properties of posture muscle in children with Spinal Muscular Atrophy.
  The biomechanical and viscoelastic properties of the posture muscle in children with Spinal Muscular Atrophy. will be measured with the MyotonPRO device.

SUMMARY:
The primary aim of the study was to measure the intra-rater and inter-rater reliability of MyotonPRO in measuring postural muscle tone and mechanical properties in individuals with spinal muscular atrophy (SMA). The secondary aim is to question the existence of a relationship between the functional levels of individuals with SMA and their muscle tone and biomechanical properties. It is assumed that the outputs to be obtained from this research will form the norm data for moyotonometer evaluation in children with SMA.

DETAILED DESCRIPTION:
It seems to be important to examine peripheral changes in the pathogenesis of SMA. Although it shows that the target center in SMA is alpha motor neurons located in the anterior horn of the spinal cord, considering the interaction network of interneurons, cerebellum, neuromuscular junction, gamma-alpha motor neuron pool, descending and ascending pathways, and reflex arc, it has potential to be investigated in individuals with SMA. This suggests that it may have important consequences for peripheral mechanisms. It may be important to examine muscle mechanical properties to reveal any potential correlations between SMA types and disease progression. In addition, moyotonometer results can be a key evaluation method in examining treatment efficacy, diagnosis and disease course. However, in order for these activities to be observed with myotonometer, first of all, the reliability of its use in individuals with SMA should be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Between 0-4 years old
* Diagnosed with spinal muscular atrophy (SMA)
* Children who continue their medical treatment at home and are not in intensive care
* Children of families who agreed to participate in the study and approved the informed consent form.

Exclusion Criteria:

* Children of families who disagreed to participate in the study

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study was to be conducted with children with a diagnosis of Spinal Muscular Atrophy (SMA) followed in the Pediatric Chest Diseases Outpatient Clinic at Bağcılar Medipol Mega University Hospital and Istanbul Medipol Hospital, and with their families meeting the inclusion criteria of the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Biomechanical and Viscoelastic Properties | Day 1.
  The biomechanical and viscoelastic properties of the plantar fascia will be measured with MyotonPRO device. The MyotonPRO (Tallin, Estonia) is a portable hand-held myotonometer. This device is non-invasive and provides a quantitative assessment of a muscle's viscoelastic properties. These properties are characterized by different parameters such as tone, elasticity, and stiffness. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Kutlutürk Yıkılmaz, Principal Investigator — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Seval Kutlutürk Yıkılmaz, Istanbul, Kavacık
  - Seval Kutlutürk Yıkılmaz, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided